CLINICAL TRIAL: NCT06297902
Title: RAdiotherapy With FDG-PET Guided Dose-PAINTing Compared With Standard Radiotherapy for Primary Head and Neck Cancer-3 Randomized, Multicentre, Phase II Trial
Brief Title: RAdiotherapy With FDG-PET Guided Dose-PAINTing Compared With Standard Radiotherapy for Primary Head and Neck Cancer-3
Acronym: RADPAINT-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Einar Dale, Senior Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023_31
Record Dates: First submitted 2024-02-12; First posted 2024-03-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Radiotherapy Side Effect
Keywords: Dose painting; 18F-FDG; Positron emission tomography; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Phase 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose painting (Experimental): Radiation dose will be escalated to the hypermetabolic part of the tumor (maximum point dose 83.3 Gy), shown in pre-treatment FDG-PET images. Dose escalation will be applied to these regions during the first half of the fractionated treatment (17 of 34 fractions).
  Interventions: Radiation: Dose painting
- Standard radiotherapy (No Intervention): Homogeneous dose to the tumor.

INTERVENTIONS:
Radiation: Dose painting — Dose painting
  Arms: Dose painting

SUMMARY:
The objective of the RADPAINT-3 trial is to investigate whether dose painting is safe compared to standard radiotherapy. RADPAINT-3 is a randomized, non-inferiority, multi-center phase II study, initiated at the Section for Head and Neck Cancer, Department of Oncology, Oslo University Hospital, accruing from first half of 2024. The primary endpoint is frequency of grade ≥ 3 (CTCAE v5.0) mucosal ulcers one year after treatment. The expected inclusion period is three years, total study duration is six years and planned inclusion number is 100 patients. The collaborating sites are St Olav´s Hospital and Haukeland University Hospital. The patients will be randomized 1:1 to either standard radiotherapy (2 Gy x 34; total dose 68 Gy) or experimental radiotherapy (dose painting). All patients will have 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission computed tomography (FDG-PET/CT) prior to radiotherapy. In the experimental arm, we will escalate the dose to the hypermetabolic part of the tumor (maximum point dose 83.3 Gy), shown in pre-treatment FDG-PET images. Dose escalation will be applied to these regions during the first half of the fractionated treatment (17 of 34 fractions). The patients in both arms will receive concomitant nimorazole (hypoxic radiosensitizer) and concomitant cisplatin if indicated according to standard treatment. The main inclusion criterion is patients with human-papillomavirus (HPV)-unrelated head and neck cancer with poor prognosis.

The RADPAINT-3 trial includes a translational sub-study where we aim to elucidate underlying mechanisms related to the radiotherapy effect, by investigating blood samples. Analysis of cytokines in repetitive blood samples may predict both tumor response and toxicity. The data derived from this sub-study, will be further explored using artificial intelligence.

If RADPAINT-3 shows that there is no excess toxicity, we will continue the study after a new protocol has been approved. The new primary endpoint will be local control at 1 year after radiotherapy. Power analysis show that we will need in total 182 evaluable patients including the 100 patients from RADPAINT-3. The translational sub-study will then be extended to investigate genetic expression data from pre-therapy routine tumor biopsies and correlate this with the analysis of blood samples and tumor control.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically verified invasive squamous cell carcinoma of the head and neck region; Sinonasal cancer, oral cavity cancer, hypopharynx cancer, larynx cancer, HPV negative oropharyngeal cancer and T4 (any N) HPV positive oropharyngeal cancer.
2. Patients planned for standard curative RT (with or without concomitant chemotherapy [cisplatin, or cetuximab], with or without nimorazole hypoxic cell radiosensitizer)
3. Age > 18 years
4. WHO performance status 0-2
5. Signed informed consent
6. Ability to understand information about the study and to complete questionnaires

Exclusion Criteria:

1. All diagnoses, cT1 cN0-N1 cM0
2. Glottic cancer cT1-T2 cN0 cM0
3. HPV positive oropharyngeal carcinoma T1-T3 (any N)
4. Diabetes mellitus
5. Use of anticoagulant medication
6. Active smoking and/or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Late mucosal ulcer | 1 year
  Presence of grade ≥ 3 mucosal ulcers (as defined by CTCAE v5.0)

SECONDARY OUTCOMES:
Early toxicity | At end of treatment - 7 weeks after inclusion
  CTCAE v5.0
Late toxicity | 1 and 3 years
  CTCAE v5.0
Odynophagia | 1 year
  EORTC QLQ-H&N43
Health-related quality of life | Up to 3 years
  EORTC QLQ-C30

OTHER OUTCOMES:
Cytokines | 1 year and 3 years
  Identify panels of cytokines measured in blood at the start of RT to predict the risk of toxicity. Blood samples will be collected before the start of treatment, after 10 Gy of radiation, at the end of therapy (7 weeks after inclusion), after 3 months of follow up (coinciding with response evaluation with FDG-PET/CT), after 1 year and fresh frozen at -80°C. Cytokine profiling will be performed by the 48-plex Luminex assay,

CONTACTS AND LOCATIONS:
Overall Officials: Einar Dale, Principal Investigator — Oslo University Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evensen ME, Furre T, Malinen E, Londalen AM, Dale E. Mucosa-sparing dose painting of head and neck cancer. Acta Oncol. 2022 Feb;61(2):141-145. doi: 10.1080/0284186X.2021.2022200. Epub 2022 Jan 6. No abstract available. PMID 34991431